CLINICAL TRIAL: NCT01186120
Title: Percutaneous Treatment of LONG Native Coronary Lesions With Drug-Eluting Stent-V:Everolimus-eluting(PROMUS-ELEMENT) vs. Biolimus A9-Eluting(NOBORI) Stents
Brief Title: Everolimus-eluting(PROMUS-ELEMENT) vs. Biolimus A9-Eluting(NOBORI) Stents for Long-Coronary Lesions
Acronym: LONG-DES-V
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Chairman,Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-0036
Record Dates: First submitted 2010-08-18; First posted 2010-08-23 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Coronary Artery Disease
Keywords: coronary disease; stent
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biolimus A9-eluting stent (Experimental): NOBORI stent
  Interventions: Device: Biolimus A9-eluting stent
- Everolimus-eluting stent (Active Comparator): PROMUS ELEMENTE stent
  Interventions: Device: Everolimus-eluting stent

INTERVENTIONS:
Device: Biolimus A9-eluting stent — drug-eluting stent
  Other Names: NOBORI stent
  Arms: Biolimus A9-eluting stent
Device: Everolimus-eluting stent — drug-eluting stent
  Other Names: PROMUS ELEMENT stent
  Arms: Everolimus-eluting stent

SUMMARY:
This randomized study is a multi-center, randomized, study to compare the efficacy of biolimus A9-eluting stent (Nobori) vs. everolimus-eluting stent (Promus Element) for long coronary lesions.

DETAILED DESCRIPTION:
Following angiography, patients with significant diameter stenosis >50% and lesion length(> 25mm) requiring single or multiple long-stent placement(total stent length 28mm) by visual estimation and eligible for LONG-DES V trial inclusion and exclusion criteria will be randomized 1:1 to a) NOBORI and b) PROMUS-ELEMENT stent by the stratified randomization method.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be at least 18 years of age.
* Significant native coronary artery stenosis (>50% by visual estimate) with lesion length of more than 25mm, which requiring single or multiple long stent placement (>=28mm)
* Patients with silent ischemia, stable or unstable angina pectoris, ad Non-ST-elevation myocardial infarction
* The patient or guardian agrees to the study protocol and the schedule of clinical and angiographic follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* Any contraindication to any of the following medications: aspirin, heparin, clopidogrel, stainless steel, contrast agents, sirolimus, or everolimus.
* An elective surgical procedure is planned that would necessitate interruption of antiplatelet drugs during the first 6 months post enrollment.
* Acute ST-segment-elevation MI or cardiogenic shock
* Terminal illness with life expectancy <1 year
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
* In-stent restenosis at target vessel (either bare metal stent or drug-eluting stent segment, non-target vessel ISR is permitted) Patients with EF<30%.
* Serum creatinine level >=3.0mg/dL or dependence on dialysis.
* Patients with left main stem stenosis (>50% by visual estimate).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2010-08; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
In-segment late luminal loss | 9 month angiographic follow-up

SECONDARY OUTCOMES:
Death (all-cause and cardiac) | 1 year
Myocardial infarction | 1 year
stent thrombosis(ARC criteria) | 1 year
target-lesion revascularization | 1 year
target-vessel revascularization | 1 year
Procedural success | at 1 day
Death (all-cause and cardiac) | one month
Death (all-cause and cardiac) | 9 months
Myocardial infarction | one month
Myocardial infarction | 9 months
Composite of death or MI | one month
Composite of death or MI | 9 months
Composite of death or MI | 1 year
Composite of cardiac death or MI | one month
Composite of cardiac death or MI | 9 months
Composite of cardiac death or MI | 1 year
target-lesion revascularization | one month
target-lesion revascularization | 9 months
target-vessel revascularization | one month
target-vessel revascularization | 9 months
stent thrombosis(ARC criteria) | one month
stent thrombosis(ARC criteria) | 9 months
In-stent late loss | 9 month angiographic follow-up
8. Target-vessel failure (death from any cause, myocardial infarction, and ischemic-driven target-vessel revascularization) | 12 months
In-stent and in-segment restenosis | 9 month angiographic follow-up
Angiographic pattern of restenosis | 9 month angiographic follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD.,PhD., Principal Investigator — Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine
Locations (11):
- South Korea (11):
  - Soonchunhyang University Hospital, Buchen, Bucheon-si
  - Soonchunhyang University Cheonan Hospital, Cheonan
  - Kangwon National University Hospital, Chooncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - NHIC Ilsan Hospital, Ilsan
  - Dong-A University Medical Center, Pusan
  - Inje University Pusan Paik Hospital, Pusan
  - Asan Medical Center, Seoul
  - Catholic University, Kangnam St. Mary's Hospital, Seoul

REFERENCES:
- [Derived] Kang DY, Jang JS, Chang M, Lee CH, Lee PH, Ahn JM, Lee SW, Kim YH, Park SW, Park DW, Park SJ; LONG-DES Investigators. Comparison of Different Types of Drug-Eluting Stents for De Novo Long Coronary Artery Lesions. JACC Asia. 2022 May 24;2(4):446-456. doi: 10.1016/j.jacasi.2022.02.009. eCollection 2022 Aug. PMID 36339368
- [Derived] Lee JY, Park DW, Kim YH, Ahn JM, Kim WJ, Kang SJ, Lee SW, Lee CW, Park SW, Yun SC, Yang TH, Lee BK, Lee NH, Yang JY, Shin WY, Park HS, Kim KS, Hur SH, Lee SY, Park JS, Choi YS, Lee SU, Her SH, Park SJ. Comparison of biolimus A9-eluting (Nobori) and everolimus-eluting (Promus Element) stents in patients with de novo native long coronary artery lesions: a randomized Long Drug-Eluting Stent V trial. Circ Cardiovasc Interv. 2014 Jun;7(3):322-9. doi: 10.1161/CIRCINTERVENTIONS.113.000841. Epub 2014 May 13. PMID 24823426